CLINICAL TRIAL: NCT03462186
Title: Promoting Patient Engagement in Clinical Preventive Services: Evaluating the Use of Healthfinder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20011992
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Invitation to use healthfinder website
  Interventions: Other: Healthfinder invitation
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Healthfinder invitation — Invitation to use healthfinder (healthfinder.gov/myhealthfinder
  Arms: Intervention

SUMMARY:
Clinical preventive services (CPS) are fundamental to early disease detection and improvement of health outcomes but are often poorly understood and utilized by patients. Myhealthfinder is a web-based tool developed by the Office of Disease Prevention and Health Promotion (https://healthfinder.gov). This study tests the "prescription" of myhealthfinder to engage patients in CPS, improve patient-clinician communication and increase uptake of CPS.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled wellness appointment with primary care provider

Exclusion Criteria:

* Inability to read English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1092 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Uptake of clinical preventive services | 3 months
  Percent up-to-datedness on cancer screening (cervical, breast, colon, lung cancer); immunizations (influenza, pneumonia) and cardiovascular disease (hypercholesterolemia, diabetes). This will be calculated based on the number of recommended services as identified on the healthfinder website based on age/gender that each patient has received within the recommended time frame.
Change in communication and health knowledge | Immediately after the intervention
  Patient survey asking about knowledge of recommended preventive services and communication with clinician; qualitative themes from audio-recordings of clinician-patient visit with subset of randomly selected patients

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Tong, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No